CLINICAL TRIAL: NCT01477866
Title: Utility Of Citogenex Administration In Patients With Colon-Rectal Cancer
Acronym: CITOGENEX PA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: the study has never started
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Manfredi Rizzo, Assistant Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CITOGENEX CRC
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- citogenex (Experimental): citogenex + conventional therapy
  Interventions: Dietary Supplement: citogenex; Other: conventional therapy
- conventional therapy (Active Comparator): conventional therapy
  Interventions: Other: conventional therapy

INTERVENTIONS:
Dietary Supplement: citogenex — CITOGENEX is a dietary supplement of insoluble polysaccharides, of Lactobacillus Casei (specific type) and of Bifidobacterium Lactis (specific type).
  Arms: citogenex
Other: conventional therapy — conventional therapy for colon-rectal cancer

SUMMARY:
The main aim of the present study is to test the efficacy and safety of CITOGENEX administration in patients with colon-rectal cancer.

DETAILED DESCRIPTION:
CITOGENEX is a dietary supplement of insoluble polysaccharides, of Lactobacillus Casei (specific type) and of Bifidobacterium Lactis (specific type). These subspecies of probiotics bacteria have been shown to be effective in improving the immunity. Several trials are currently underway, in order to evaluate the effects of probiotics as potential novel therapies in addition to traditional therapeutic approaches. Although probiotics do not play an anti-tumor action per se, these agents may significantly contribute to decrease the typical side effects due to traditional anti-tumor treatments, such as gastrointestinal symptoms, immunity deficit, as well as the alterations in the gut lymphoid tissue.

It is therefore expected that CITOGENEX may have several significant beneficial effects in patients under anti-tumor treatments. In order to test this hypothesis, we will perform a randomized, single-blind, two-arms, prospective study in patients with colon-rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* stage IIIa-IIIc (AJCC/TNM)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Tomasello, MD, Study Director — University of Palermo; Francesco Cappello, MD, Study Chair — University of Palermo; Provvidenza Damiani, MD, Principal Investigator — University of Palermo; Manfredi Rizzo, MD, Principal Investigator — University of Palermo
Locations (1):
- University of Palermo, Palermo, PA, Italy